CLINICAL TRIAL: NCT06683144
Title: Effects of Feedback, Education, and Social Media Interventions Based on the Health Belief Model on Preventive Beliefs in Adults Exposed to Secondhand Smoke At Home.
Brief Title: Effects of Health Belief Model Interventions on Preventive Beliefs in Secondhand Smoke Exposure
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Ercan Asi, Research Assistant, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AU-NF-EA-01
Record Dates: First submitted 2024-11-08; First posted 2024-11-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2024-11

CONDITIONS: Secondhand Smoke Exposure
Keywords: secondhand smoke; exposure; health belief model

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Exposure feedback group (Experimental)
  Interventions: Behavioral: Exposure feedback
- Interactive education group (Experimental)
  Interventions: Behavioral: Exposure feedback; Behavioral: Interactive education
- Social media group (Experimental)
  Interventions: Behavioral: Exposure feedback; Behavioral: Social media post

INTERVENTIONS:
Behavioral: Exposure feedback — * Determining the actual SHS exposure risk level and providing feedback.
  * Determining the urinary cotinine test result and providing feedback.
  * Feedback on the consistency or difference between the perceived SHS exposure risk level and the actual SHS exposure risk level.
Behavioral: Interactive education — Slide presentation, video presentation, Q&A, evaluation of learning and discussion of results
  Arms: Interactive education group
Behavioral: Social media post — Sharing informational materials such as messages, brochures, and videos related to SHS exposure, including ways to protect yourself from SHS exposure and the adverse health effects of SHS exposure.
  Arms: Social media group

SUMMARY:
The aim of this study was to compare the effects of feedback, interactive education, and social media interventions based on the health belief model on protective beliefs in adults at risk of exposure to secondhand smoke at home.

DETAILED DESCRIPTION:
Secondhand smoke (SHS) exposure, also known as environmental tobacco smoke, passive smoke or involuntary smoke, is caused by the burning of cigarettes and other tobacco products and the smoke exhaled by a smoker. Although Turkey is one of the best countries in combating SHS exposure, one in four adults is exposed to SHS at home. One of the most important reasons for this exposure is the lack of deterrent policies for the home environment, which is considered a private area. It is entirely possible for non-smoking individuals to be protected from SHS exposure at home through their own efforts. In this context, the knowledge, behaviors and perceptions of non-smoking adults about exposure are important in preventing or reducing SHS exposure at home. Interventions based on the behavior change model can be effective in developing protective behaviors in adults at risk of SHS exposure at home. Individual and group interventions using multiple educational materials and methods based on the Health Belief Model (HBM) (SHS exposure feedback, interactive group education and social media sharing) can develop protective behaviors in individuals at home.

ELIGIBILITY:
İnclusion Criteria

* Non-smokers aged 18-64 who live with at least one smoker,
* Literate individuals,
* Individuals who own a smartphone,
* Individuals who voluntarily agree to participate in the study.

Exclusion Criteria:

* Individuals who do not speak Turkish,
* Pregnant individuals,
* Participants who have been living apart from SHS exposure sources in the week leading up to data collection.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 93 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-06-10 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
Health belief model scale for prevention behaviors of secondhand smoke exposure (HBM-SHS) | Baseline and at first month later after intervention
  The 35-item scale, scored on a five-point Likert scale from "Strongly Disagree (1)" to "Strongly Agree (5)," assesses six subdimensions: "perceived susceptibility," "perceived seriousness," "perceived benefits," "perceived barriers," "self-efficacy," and "behavioral cues." Items on "perceived susceptibility" and "perceived barriers" are reverse coded. Scores range from 35 to 175, with higher scores indicating stronger health beliefs about SHS exposure and greater beliefs in each subdimension.

SECONDARY OUTCOMES:
Secondhand Smoke Exposure Risk Assessment | Baseline and at first month later after intervention
  Risk assessment is conducted through four questions addressing whether there is a smoker in the household, household tobacco use rules, tobacco use in enclosed areas, and the time since the last use. Responses are scored categorically: absence of risk is scored as 0, while the presence and intensity of risk are scored as 1 or more. A score of at least one indicates "risk." SHS exposure risk is scored from 0 to 10, with any score of 1 or above indicating the presence of risk. Total risk assessment scores are represented on a real risk scale of 0-10. According to expert evaluations, the content validity index (CVI) of the questions assessing participants' SHS exposure risk level is 0.86.
Actual Risk Assessment | Baseline and at first month later after intervention
  In adults at risk of SHS exposure, urinary cotinine analysis will be conducted using a cotinine urine test kit. The test detects cotinine in the urine, indicating SHS exposure. The strip is dipped into the urine sample for 10 seconds, and the result is read within 5 minutes. In a negative result, both the control (C) and test (T) lines will appear, while in a positive result, only the control line (C) will appear. If neither the C nor T lines are visible, or if only the T line appears, the test is invalid.
Perceived SHS Exposure Risk | Baseline and at first month later after intervention
  In adults, SHS exposure risk will be assessed based on the perceived level of risk. Participants' awareness of SHS exposure will be measured by their responses to the question, "How would you describe your risk of being exposed to SHS in your home?" with options such as "No risk at all," "Somewhat at risk," or "At very high risk." Additionally, participants' perceived SHS exposure risk level will be evaluated based on their numerical responses to the question, "What would your risk of SHS exposure in your home be on a scale from 0 to 10?" Each number will represent the participant's perceived (exposure risk probability) risk.
ThirdHand Smoke Beliefs Scale (BATHS) | Baseline and at first month later after intervention
  This scale was developed by Haardörfer and colleagues in 2017 to identify beliefs about third-hand smoke (THS). The scale includes 5 items related to the health effects of THS and 4 items regarding its persistence in the environment. The items are rated using a 5-point Likert scale, with the following coding: 5 = Strongly agree, 4 = Agree, 3 = Neutral, 2 = Disagree, 1 = Strongly disagree. The total score of the scale is obtained by dividing the sum of the item scores by the number of items. A score closer to 5 for each item indicates the individual believes in the health and environmental effects of THS, while a score closer to 1 indicates disbelief.

CONTACTS AND LOCATIONS:
Locations (1):
- Akdeniz University Faculty of Nursing, Antalya, Konyaaltı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No